CLINICAL TRIAL: NCT03646227
Title: Multi-Drug Resistant Organism Network - MDRO Network
Brief Title: Multi-Drug Resistant Organism Network
Acronym: MDRO Network
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00071149; UM1AI104681 (NIH)
Record Dates: First submitted 2018-08-15; First posted 2018-08-24 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Infections Resistant to Multiple Drugs; Bacterial Infections
Keywords: Carbapenem-resistant enterobacteriaceae (CRE); Carbapenem-resistant Pseudomonas aeruginosa (CRPA); Klebsiella pneumoniae; Acinetobacter baumannii (CRAb); Bloodstream infection (BSI); Microbiological characterization
MeSH Terms: conditions — Bacterial Infections; Sepsis | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A sample of all MDRO isolates (bacterial isolates) will be sent to a central research laboratory for molecular and microbiological characterization. In addition, antimicrobial susceptibility testing, determination of mechanisms of antibiotic resistance, and strain typing will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard of Care — There is no prescribed intervention for this study. Standard of care will be captured in the eCRF.

SUMMARY:
This study is specifically designed to provide observational data which can be used to help in the design of future randomized clinical trials on both therapeutics and diagnostics for MDRO infections. To this end, clinical and epidemiological data will be collected on patients who have MDRO isolated from clinical cultures during hospitalization, as well as descriptions of the outcomes of patients treated with various antimicrobial regimens. Molecular and microbiological characterization will also be performed on MDRO isolates. These data will include a detailed clinical and epidemiological description of patients including identifying potential barriers to enrollment in future trials. In addition, data will be collected on species, strain type, and mechanism of drug resistance of the causative organism. Knowing the molecular characteristics will further inform future trial design as not all diagnostics detect and not all therapeutics are active against the same mechanisms of resistance.

DETAILED DESCRIPTION:
This is a prospective multi-center study. At each hospital, study personnel will screen the microbiology laboratory logs to identify all patients found to have a MDRO isolate from one or more anatomical sites during hospitalization. For each patient identified, designated site personnel will access the patient's medical record and use web-based data entry to enter the relevant data into the electronic case report form (eCRF) in the study's centralized database.

A sample of all MDRO isolates (bacterial isolates) will be sent to a central research laboratory for molecular analysis which will include strain typing. In addition, the mechanism of resistance will be determined by performing PCR and/or Whole Genome Sequencing.

Aim 1. Identification of target population and high volume centers. The prevalence of specific MDRO is extremely variable in various patient populations. In addition, over time, prevalence patterns for specific MDRO tend to change. The data collection carried out under this protocol will provide real-time data on which patients are the target population for any trial directed against MDRO infection. Also, the data collected will indicate which geographic areas and which centers have the highest incidence of MDRO infections. This will facilitate rational site selection for future trials.

Aim 2. Provide data on impact of potential inclusion/exclusion criteria on enrollment in future trials.

Detailed clinical data will be collected to guide the future development of clinical trials. The eCRF is designed to collect data on the most common barriers to enrollment in clinical trials. Data can then be used in the design of future trials to be presented to pharmaceutical companies, as well as to regulators from the FDA, to provide a rationale for requesting exceptions in inclusion/exclusion criteria. This will result in clinical trials that are more readily generalizable.

Aim 3. Provide data on expected outcomes of patients with MDRO infections for power and sample size calculations for future trials.

In the MDRO network, detailed outcomes data will be collected. Data will include survival and microbiologic clearance outcomes when available. In addition, anatomical site specific clinical symptomatic outcomes, modeled on FDA guidance documents, will be documented. Data obtained will aid in guiding the design of future clinical trials by providing data needed for power and sample size calculations.

All hospitalized patients, including pediatric patients, who have an MDRO isolated from a clinical culture will be included. Patients who have a positive culture for MDRO that is obtained outside the hospital setting will not be included, to ensure the ability to collect MDRO isolates and sufficient clinical data. Overall enrollment is expected to be 7000.

This study will request a waiver of informed consent, consistent with CFR Title 45 part 46.116(d). The study does not involve direct interaction with human subjects. The medical records of patients admitted to the hospital will be screened and data collected from those records according this protocol. The patients will not be approached to obtain information, no intervention is being tested. MDRO isolates will be obtained from existing standard of care microbial testing.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients.
* Must have at least one multi-drug resistant organism isolated from a clinical culture while hospitalized.

Exclusion Criteria:

* Patients who do not have a positive culture during hospitalization.
* Patients who's only positive culture was obtained outside of hospital admission.
* Patients who have cystic fibrosis and a CRPa infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohorts will be constructed for each MDRO of eligible patients by investigating hospitalized patients who have an MDRO isolated in clinical cultures from any anatomical site. This study will be conducted under a waiver of informed consent to facilitate universal inclusion. All patients who are admitted to one of the participating hospitals and who have an MDRO - as defined in the specific sub-study protocol (Appendices) - isolated in a clinical culture are targeted for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 6496 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Disposition at Discharge | Up to 1 year from index culture date
  The disposition at discharge is a composite of different locations, to which the subject is discharged (skilled nursing facility, home, long term acute care facility, transfer to another hospital, death, or hospice) and it is used to compare patient outcomes based on MDRO collected form the subject.
Charlson Score | At 90 days after discharge from the index hospitalization
  Components of the Charlson Score are collected from the medical record and the Charlson comorbidity index is calculated to determine chronically ill subjects.
Pitt Bacteremia Score | On the day of index culture
  Components of the Pitt Bacteremia Score are collected from the medical record and the Pitt bacteremia score is calculated to determine acutely ill subjects.
Source of positive culture | At collection of the MDRO isolates
  The differences in outcomes based on the anatomic source of the positive culture are determined. The anatomic sources collected are blood, respiratory, urine, wound, abdominal, and other, which is collected from the medical record.
Length of Stay | Up to 1 year from index culture date
  The length of stay is determined by the hospital admission and discharge dates, which is collected from the medical record.
ICU Admissions | Up to 1 year from index culture date
  The total number ICU days during the index hospitalization will be collected from the medical record to determine high risk populations and exposure.
Antibiotic Summary | Only during hospitalization and up to one year from index culture date
  All antibiotics administered during the hospital stay will be collected from the medical record. The antibiotic name, duration of therapy, frequency of dosing, dosage, and reason for discontinuation will be collected for the antibiotics of interest.
Survival Status | 90 days from discharge or up to one year from index hospitalization.
  Survival status will be collected through 90 days after discharge from index hospitalization, up to one year, to determine mortality.
Readmission Status | 90 days after discharge from index hospitalization.
  Readmission data will be collected through 90 days after discharge from index hospitalization to determine readmission.

CONTACTS AND LOCATIONS:
Overall Officials: David van Duin, MD. PhD, Principal Investigator — University of North Carolina; Robert Bonomo, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (4):
- Duke Clinical Research Institute, Durham, North Carolina, United States
- The University of Queensland Centre for Clinical Research, Herston, Queensland, Australia
- Huashan Hospital, Shanghai, Shanghai Municipality, China
- Universidad El Bosque, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Yes
The resulting SAP and results will be shared and discussed within the MDRO Publications Committee for the purpose of manuscript developing, and to inform the design of future clinical trials.
Supporting Information: Study Protocol, SAP
Time Frame: Starting January 2017 through November 2019
Access Criteria: Must have an executed CDA and sub-award with ARLG/Duke for this specific purpose.

REFERENCES:
- [Background] Clatworthy AE, Pierson E, Hung DT. Targeting virulence: a new paradigm for antimicrobial therapy. Nat Chem Biol. 2007 Sep;3(9):541-8. doi: 10.1038/nchembio.2007.24. PMID 17710100
- [Background] Infectious Diseases Society of America (IDSA); Spellberg B, Blaser M, Guidos RJ, Boucher HW, Bradley JS, Eisenstein BI, Gerding D, Lynfield R, Reller LB, Rex J, Schwartz D, Septimus E, Tenover FC, Gilbert DN. Combating antimicrobial resistance: policy recommendations to save lives. Clin Infect Dis. 2011 May;52 Suppl 5(Suppl 5):S397-428. doi: 10.1093/cid/cir153. No abstract available. PMID 21474585
- [Background] Vardakas KZ, Rafailidis PI, Konstantelias AA, Falagas ME. Predictors of mortality in patients with infections due to multi-drug resistant Gram negative bacteria: the study, the patient, the bug or the drug? J Infect. 2013 May;66(5):401-14. doi: 10.1016/j.jinf.2012.10.028. Epub 2012 Nov 6. PMID 23142195
- [Background] Zasowski EJ, Rybak JM, Rybak MJ. The beta-Lactams Strike Back: Ceftazidime-Avibactam. Pharmacotherapy. 2015 Aug;35(8):755-70. doi: 10.1002/phar.1622. PMID 26289307
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] van Duin D, Perez F, Rudin SD, Cober E, Hanrahan J, Ziegler J, Webber R, Fox J, Mason P, Richter SS, Cline M, Hall GS, Kaye KS, Jacobs MR, Kalayjian RC, Salata RA, Segre JA, Conlan S, Evans S, Fowler VG Jr, Bonomo RA. Surveillance of carbapenem-resistant Klebsiella pneumoniae: tracking molecular epidemiology and outcomes through a regional network. Antimicrob Agents Chemother. 2014 Jul;58(7):4035-41. doi: 10.1128/AAC.02636-14. Epub 2014 May 5. PMID 24798270
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Background] Chow JW, Yu VL. Combination antibiotic therapy versus monotherapy for gram-negative bacteraemia: a commentary. Int J Antimicrob Agents. 1999 Jan;11(1):7-12. doi: 10.1016/s0924-8579(98)00060-0. PMID 10075272
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Derived] Jiang J, Komarow L, Hill C, Boutzoukas AE, Hanson B, Arias CA, Bonomo RA, Evans S, Doi Y, Satlin MJ, Weston G, Cober E, Valderrama-Beltran SL, Mendoza SS, Liu Z, Fries BC, Tambyah PA, Chambers HF, Fowler VG Jr, van Duin D, Kreiswirth BN, Chen L. Molecular Epidemiology and Clinical Characterization of Carbapenemase-Producing Enterobacter Species From an International Cohort. J Infect Dis. 2025 Jul 11;231(6):1489-1501. doi: 10.1093/infdis/jiae616. PMID 39667036
- [Derived] Boutzoukas AE, Mackow N, Giri A, Komarow L, Hill C, Chen L, Doi Y, Satlin MJ, Arias C, Wang M, Mora Moreo L, Herc E, Cober E, Weston G, Patel R, Bonomo RA, Fowler V, van Duin D. Increased mortality in hospital- compared to community-onset carbapenem-resistant enterobacterales infections. J Antimicrob Chemother. 2024 Nov 4;79(11):2916-2922. doi: 10.1093/jac/dkae306. PMID 39236214
- [Derived] Wang M, Ge L, Chen L, Komarow L, Hanson B, Reyes J, Cober E, Alenazi T, Zong Z, Xie Q, Liu Z, Li L, Yu Y, Gao H, Kanj SS, Figueroa J, Herc E, Cordova E, Weston G, Ananth Tambyah P, Garcia-Diaz J, Kaye KS, Dhar S, Munita JM, Salata RA, Vilchez S, Stryjewski ME, Villegas Botero MV, Iovleva A, Evans SR, Baum K, Hill C, Kreiswirth BN, Patel R, Paterson DL, Arias CA, Bonomo RA, Chambers HF, Fowler VG Jr, Satlin MJ, van Duin D, Doi Y; Multi-Drug Resistant Organism Network Investigators. Clinical Outcomes and Bacterial Characteristics of Carbapenem-resistant Acinetobacter baumannii Among Patients From Different Global Regions. Clin Infect Dis. 2024 Feb 17;78(2):248-258. doi: 10.1093/cid/ciad556. PMID 37738153
- [Derived] Wang M, Earley M, Chen L, Hanson BM, Yu Y, Liu Z, Salcedo S, Cober E, Li L, Kanj SS, Gao H, Munita JM, Ordonez K, Weston G, Satlin MJ, Valderrama-Beltran SL, Marimuthu K, Stryjewski ME, Komarow L, Luterbach C, Marshall SH, Rudin SD, Manca C, Paterson DL, Reyes J, Villegas MV, Evans S, Hill C, Arias R, Baum K, Fries BC, Doi Y, Patel R, Kreiswirth BN, Bonomo RA, Chambers HF, Fowler VG Jr, Arias CA, van Duin D; Multi-Drug Resistant Organism Network Investigators. Clinical outcomes and bacterial characteristics of carbapenem-resistant Klebsiella pneumoniae complex among patients from different global regions (CRACKLE-2): a prospective, multicentre, cohort study. Lancet Infect Dis. 2022 Mar;22(3):401-412. doi: 10.1016/S1473-3099(21)00399-6. Epub 2021 Nov 9. PMID 34767753
- [Derived] van Duin D, Arias CA, Komarow L, Chen L, Hanson BM, Weston G, Cober E, Garner OB, Jacob JT, Satlin MJ, Fries BC, Garcia-Diaz J, Doi Y, Dhar S, Kaye KS, Earley M, Hujer AM, Hujer KM, Domitrovic TN, Shropshire WC, Dinh A, Manca C, Luterbach CL, Wang M, Paterson DL, Banerjee R, Patel R, Evans S, Hill C, Arias R, Chambers HF, Fowler VG Jr, Kreiswirth BN, Bonomo RA; Multi-Drug Resistant Organism Network Investigators. Molecular and clinical epidemiology of carbapenem-resistant Enterobacterales in the USA (CRACKLE-2): a prospective cohort study. Lancet Infect Dis. 2020 Jun;20(6):731-741. doi: 10.1016/S1473-3099(19)30755-8. Epub 2020 Mar 6. PMID 32151332
- See also: Antibacterial Resistance Leadership Group (ARLG) — http://www.arlg.org

DOCUMENTS (2):
  • Study Protocol (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT03646227/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT03646227/SAP_001.pdf